CLINICAL TRIAL: NCT03378284
Title: A Randomized, Open-label, Active-controlled, Multiple Dose Phase 1 Clinical Trial to Evaluate Safety, Tolerability, and Pharmacodynamics of Tegoprazan After Oral Administration in Healthy Male Volunteers
Brief Title: A Study to Evaluate Safety, Tolerability, and PD of Tegoprazan on Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_APA_108
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2017-12

CONDITIONS: Pharmacodynamics; Healthy Male Volunteers
MeSH Terms: interventions — tegoprazan; YH 1885

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tegoprazan(Test drug) (Experimental): Tegoprazan drug QD for 7 days
  Interventions: Drug: Tegoprazan
- Active comparator drug (Active Comparator): Active comparator drug QD for 7 days
  Interventions: Drug: Revaprazan

INTERVENTIONS:
Drug: Tegoprazan — Tegoprazan QD for 7 days
  Arms: Tegoprazan(Test drug)
Drug: Revaprazan — Revaprazan QD for 7 days
  Arms: Active comparator drug

SUMMARY:
A randomized, open-label, active-controlled, multiple dose phase 1 clinical trial to evaluate safety, tolerability, and pharmacodynamics of tegoprazan after oral administration in healthy male volunteers

DETAILED DESCRIPTION:
* To compare the pharmacodynamics of multiple oral dose of tegoprazan versus the pharmacodynamics of multiple oral dose of comparator drug in healthy male volunteers.
* To evaluate the safety and tolerability of multiple oral dose of tegoprazan in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged ≥ 19 years and ≤ 50 years
* Body weight of ≥ 55.0 kg and ≤ 90.0 kg, with body mass index (BMI) of ≥ 18.0 kg/m2 and ≤ 27.0 kg/m2 at the time of screening

Exclusion Criteria:

* Presence or history of clinically significant diseases
* Presence or history of gastrointestinal disorder (gastric ulcer, GERD, Crohn's disease, etc.)
* Hypersensitivity to drugs containing study drug or proton pump inhibitor and other drugs (aspirin, antibiotics, etc.) or history of clinically significant hypersensitivity
* Serologic test positive
* Abnormal obstacle to insertion and maintenance of pH meter catheter
* History of drug abuse
* Excessive caffeine intake or persistent alcohol intake
* Not use of a medically acceptable method of contraception

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
Gastric pH | up to 7 days
  Gastric pH
Serum gastrin concentration | up to 9 days
  Serum gastrin concentration

CONTACTS AND LOCATIONS:
Overall Officials: In Jin Jang, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided